CLINICAL TRIAL: NCT06128226
Title: A Multicenter Selective Screening Study to Investigate the Frequency of Neuronal Ceroid Lipofuxinosis Type 2 (CLN2) in the Presence of Nonspecific Neurological Findings Accompanying Seizures Between the Ages of 2 and 6
Brief Title: A Multicenter Selective Screening Study to Investigate the Frequency of Neuronal Ceroid Lipofuxinosis Type 2 (CLN2)
Acronym: ENIGMA
Status: Recruiting | Type: Observational
Sponsor: Nadir Hastalıkları Araştırma Derneği (Other)
Responsible Party: Sponsor
Other Study IDs: K-AO003-ENIGMA
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Neuronal Ceroid Lipofuxinosis Type2 (CLN2)
Keywords: Neuronal; Genetics; Metabolism; Rare
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For Tripeptidyl Peptidase 1 enzyme level measurement, blood will be taken from the patient into a 5 mL EDTA tube at Gazi University Faculty of Medicine, Metabolism Laboratory, and for patients with low enzyme activity, the genetic evaluation test will be performed with whole blood at the Gene2Info Laboratory.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Blood Sampling — For Tripeptidyl Peptidase 1 enzyme level measurement, blood will be taken from the patient into a 5 mL EDTA tube at Gazi University Faculty of Medicine, Metabolism Laboratory, and for patients with low enzyme activity, the genetic evaluation test will be performed with whole blood at the Gene2Info Laboratory.

SUMMARY:
This study is a multicenter, non-drug screening study. Enrollment period is 12 months. There are no IMP to be followed or used in the study. Patients who applied to Pediatric Metabolism, Pediatric Neurology and Developmental Pediatrics clinics with the symptoms or findings defined in the protocol as below for 12 months will be included in the study.

Children between the ages of 2 and 6, without hypoxic ischemic encephalopathy, head trauma and developmental brain anomalies, who are admitted to the Pediatric Metabolism, Pediatric Neurology and Developmental Pediatrics clinics with non-specific neurological symptoms such as idiopathic seizures of unknown etiology, speech disorders and motor dysfunctions, will constitute the target population of the study.

DETAILED DESCRIPTION:
Demographic data, medical history and family history of the patients included in the study will be recorded at their first admission. In addition, seizure frequency; cognitive functions, including assessments of language development; physical examination information including assessments of muscle strength, gait, and coordination; Data on neurological evaluation results and visual ability evaluations, such as Electroencephalography (EEG) and Magnetic Resonance Imaging (MRI), will be collected. Following the above screenings, patients between the ages of 2-6 who show at least one of the following: speech disorder with idiopathic seizures/regression in acquired speech skills, symptoms of gait and movement disorders, or photoparoxysmal response to EEG with low-frequency IFS, cerebral atrophy or preventive white matter hyperintensity on MRI, Enzyme analysis and genetic tests will be performed on children to investigate CLN2 disease.The tests are written in detail below.

For Tripeptidyl Peptidase 1 enzyme level measurement, blood will be taken from the patient into a 5 mL EDTA tube at Gazi University Faculty of Medicine, Metabolism Laboratory, and for patients with low enzyme activity, the genetic evaluation test will be performed with whole blood at the Gene2Info Laboratory.

Study endpoints are to determine the frequency of type 2 (CLN2) disease and to determine the demographic and clinical characteristics of these patients with neuronal ceroid lipofuscinosis who showed at least one of the following: speech impairment with idiopathic seizures/decline in acquired speech skills, symptoms of gait and movement disorders, or photoparoxysmal response to EEG with low-frequency IFS, cerebral atrophy or pretricular white matter hyperintensity on MRI.

ELIGIBILITY:
Inclusion Criteria:

* Girls and boys aged 6 years old
* Having a history of at least one seizure
* With a history of idiopathic seizures;

  * Speech disorder or regression in acquired speaking skills,
  * Motor dysfunctions,
  * Photoparoxysmal response to EEG with low-frequency IFS,
  * Observation of at least one of the symptoms or signs of cerebral atrophy or preventive white matter hyperintensity on MRI
* Without hypoxic ischemic encephalopathy, head trauma and developmental brain anomalies
* Not having been previously diagnosed with CLN2
* The patient and/or his/her legal representative must be willing to sign the written consent form.

Exclusion Criteria:

* Patients younger than 2 years and older than 6 years
* Patients with a known or diagnosed neurodegenerative disorder
* Patients for whom written consent form cannot be obtained from their legal representative

Ages: 2 Years to 6 Years | Sex: All
Age Groups: Child
Study Population: Children between the ages of 2 and 6, without hypoxic ischemic encephalopathy, head trauma and developmental brain anomalies, who are admitted to the Pediatric Metabolism, Pediatric Neurology and Developmental Pediatrics clinics with non-specific neurological symptoms such as idiopathic seizures of unknown etiology, speech disorders and motor dysfunctions, will constitute the target population of the study.
Sampling Method: Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Disease Frequency | 1 year
  To determine the frequency of Neuronal Ceroid Lipofuxinosis type 2 (CLN2) disease and to determine the demographic and clinical characteristics of these patients.

CONTACTS AND LOCATIONS:
Locations (34):
- Turkey (Türkiye) (34):
  - Adana City Hospital, Pediatric Metabolism, Adana
  - Adana City Hospital, Pediatric Neurology, Adana
  - Adana Medical Park Hospital, Pediatric Neurology, Adana
  - Adana Şehir Hastanesi, Developmental Pediatrics, Adana
  - Başkent University School of Medicine, petiatric Metabolism, Adana
  - Seyhan State Hospital, Pediatric Neurology, Adana
  - Çukurova University School of Medicine, Pediatric Metabolism, Adana
  - Çukurova University School of Medicine, Pediatric Neurology, Adana
  - Batman Medical Point Hospital, Pediatric Neurology, Batman
  - Batman Training and Research Hospital, Pediatric Neurology, Batman
  - Dicle University School of Medicine, Pediatric Neurology, Diyarbakır
  - Diyarbakır Gazi Yaşargil Training and Research Hospital, Developmental Pediatrics, Diyarbakır
  - Diyarbakır Gazi Yaşargil Training and Research Hospital, Pediatric Neurology, Diyarbakır
  - Elazığ Fethi Tekin City Hospital, Elâzığ
  - Fırat University School of Medicine, Pediatric Metabolism, Elâzığ
  - Gaziantep Cengiz Göçek Child's Hospital, Developmental Pediatrics, Gaziantep
  - Gaziantep Cengiz Göçek Child's Hospital, Pediatric Metabolism, Gaziantep
  - Gaziantep Cengiz Göçek Child's Hospital, Pediatric Neurology, Gaziantep
  - Gaziantep University School of Medicine, Pediatric Neurology, Gaziantep
  - Hatay Training and Research Hospital, Pediatric Neurology, Hatay
  - Necip Fazıl City Hospital, Pediatric Neurology, Kahramanmaraş
  - Sütçü İmam University School of Medicine, Pediatric Neurology, Kahramanmaraş
  - Malatya İnönü University School of Medicine, Developmental Pediatrics, Malatya
  - Malatya İnönü University School of Medicine, Pediatric Neurology, Malatya
  - Malatya Training and Reserach Hospital, Pediatric Neurology, Malatya
  - Mardin Artuklu University School of Medicine, Pediartic Endocrinology, Mardin
  - Mardin Artuklu University School of Medicine, Pediatric Neurology, Mardin
  - Mersin City Hospital, Pediatric Metabolism, Mersin
  - Mersin City Hospital, Pediatric Neurology, Mersin
  - Mersin City Hospital, Mersin
  - Mersin University School of Medicine, Pediatric eurology, Mersin
  - Şanluurfa Harran University School of Medicine, Pediatric Metabolism, Sanliurfa
  - Şanlıurfa Training and Research Hospital, Pediatric Neurology, Sanliurfa
  - Van Regional Training and Research Hospital, Van

IPD SHARING:
Plan to Share IPD: No